CLINICAL TRIAL: NCT02517931
Title: Sphenopalatine Ganglion Block for Treatment of Postdural Puncture Headache in the Emergency Department: A Prospective, Randomized, Double-Blind Placebo Controlled Study
Brief Title: Sphenopalatine Ganglion Block for Postdural Puncture Headache in the Emergency Department
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding for the project
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 204502
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sphenopalatine Ganglion Block (Active Comparator): Subjects will be asked to blow out each nostril. They will then be laid supine with a small shoulder roll and intranasal phenylephrine 0.25% (RhinallⓇ) will be sprayed once into each nostril to preemptively minimize bleeding. Sphenopalatine ganglion block will be performed by inserting long cotton tipped applicators saturated in 2% viscous lidocaine into nostril until properly seated in the posterior nasopharynx. These will be left in place for 10 minutes and then 1 mililiter of 0.5% bupivacaine will be administered down the plastic hollow shaft of each applicator via an 18g angiocatheter. The applicators will remain in place for 10 more minutes and then be removed.
  Interventions: Procedure: Sphenopalatine Ganglion Block
- Placebo (Placebo Comparator): Subjects will be asked to blow out each nostril. They will then be laid supine with a small shoulder roll and intranasal phenylephrine 0.25% (RhinallⓇ) will be sprayed once into each nostril to preemptively minimize bleeding. SPGB will be performed by inserting long cotton tipped applicators saturated in carboxymethylcellulose based lubricant (i.e. K-Y Jelly®) into nostril until properly seated in the posterior nasopharynx. These will be left in place for 10 minutes and then 1 mililiter of normal saline will be administered down the plastic hollow shaft of each applicator via an 18g angiocatheter. The applicators will remain in place for 10 more minutes and then be removed.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block — Subjects will be asked to blow out each nostril. They will then be laid supine with a small shoulder roll and intranasal phenylephrine 0.25% (RhinallⓇ) will be sprayed once into each nostril to preemptively minimize bleeding. SPGB will be performed by inserting long cotton tipped applicators saturated in 2% viscous lidocaine into nostril until properly seated in the posterior nasopharynx. These will be left in place for 10 minutes and then 1mL of 0.5% bupivacaine will be administered down the plastic hollow shaft of each applicator via an 18g angiocatheter. The applicators will remain in place for 10 more minutes and then be removed.
  Arms: Sphenopalatine Ganglion Block
Procedure: Placebo — Subjects will be asked to blow out each nostril. They will then be laid supine with a small shoulder roll and intranasal phenylephrine 0.25% (RhinallⓇ) will be sprayed once into each nostril to preemptively minimize bleeding. SPGB will be performed by inserting long cotton tipped applicators saturated in carboxymethylcellulose based lubricant (i.e. K-Y Jelly®) into nostril until properly seated in the posterior nasopharynx. These will be left in place for 10 minutes and then 1 mililiter of normal saline will be administered down the plastic hollow shaft of each applicator via an 18g angiocatheter. The applicators will remain in place for 10 more minutes and then be removed.
  Arms: Placebo

SUMMARY:
This study evaluates sphenopalatine ganglion block (SPGB) for the treatment of postdural puncture headache (PDPH) in the emergency department (ED). Half of the patients will receive a true nerve block with lidocaine and bupivacaine. The other half will receive a placebo nerve block.

DETAILED DESCRIPTION:
Postdural puncture headaches (PDPH) are a common consequence of diagnostic lumbar puncture. The gold standard treatment for a PDPH is currently an autologous epidural blood patch (AEBP), which involves placing a needle into the epidural space of the spine and then injecting 20 ml of the patients own blood through the needle and into the epidural space to form a clot over the tear in the tissue layer that causes the headache. This is an invasive procedure that carries risks of pain, bleeding, infection, and in rare cases, neurological complications. We want to test the efficacy of using a less invasive procedure, called a sphenopalatine ganglion block (SPGB), for treatment of PDPH. SPGB has been used for many years in the treatment of migraines and cluster headaches, and there are several case reports of its use to successfully treat PDPH as well. SPGB simply involves applying a local anesthetic to the mucosa in the back of each nostril to numb the nerves that cause the headache. We hope that the SPGB will reduce the number of PDPH patients that require an AEBP.

ELIGIBILITY:
Inclusion Criteria:

* Active postdural puncture headache within 7 days after diagnostic lumbar puncture
* Age ≥ 18 years.
* American Society of Anesthesiologists (ASA) physical status ≤ 3

Exclusion Criteria:

* Known coagulopathy
* Known nasal septal deviation or abnormalities
* Medical conditions contraindicated to lidocaine or bupivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Pain level with Verbal Rating Scale | 5 days
  Patients will be asked to self rate their pain with 0 as no pain at all up to 10 being the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Carly Eastin, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States